CLINICAL TRIAL: NCT00216190
Title: A Phase 4, Randomized, Double-Blind, Multi-Center, Comparator Study Evaluating the Safety and Efficacy of Dexmedetomidine Compared to IV Midazolam in ICU Subjects Requiring Greater Than Twenty-Four Hours of Continuous Sedation
Brief Title: A Safety and Efficacy Study of Dexmedetomidine in ICU Patients Requiring Continuous Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-001
Record Dates: First submitted 2005-08-31; First posted 2005-09-22 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Mechanically Ventilated and Intubated Subjects
Keywords: Sedation, ICU, Anesthesia, Dexmedetomidine, Midazolam
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine HCL Injection
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam Injection

INTERVENTIONS:
Drug: Dexmedetomidine HCL Injection
  Arms: Dexmedetomidine
Drug: Midazolam Injection
  Arms: Midazolam

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of dexmedetomidine in ICU subjects who are initially intubated, mechanically ventilated and require sedation for beyond 24 hours.

DETAILED DESCRIPTION:
Traditional agents such benzodiazepines and propofol have long been used to sedate critically ill patients. Unfortunately, these agents have serious disadvantages that may have a negative impact on patient outcomes. These disadvantages include respiratory depression, prolonged mechanical ventilation, paradoxical agitation, myocardial depression, hypotension, tachyphylaxis, physical dependence, and an unpredictable duration of action following long term infusions. Additionally, concomitant use of an opioid or other analgesic is often required for ICU patients to achieve adequate levels of pain relief, which may also prolong awakening and possibly increase respiratory depression.

Dexmedetomidine may offer a new treatment option that remedies many of the deficiencies of traditional sedatives. This agent would provide for accurate, titratable sedation and analgesia without the concurrent respiratory depression and accumulation common to other agents. It may permit greater patient interaction due to reduced impairment of cognition and may reduce risks associated with opioids due to its analgesia sparing property. Although such a drug may have important benefits for ICU patients requiring sedation for greater than 24 hours, dexmedetomidine is not currently approved for such long-term usage.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. If female, subject is non-lactating, and is either:

   1. Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
   2. Of childbearing potential but is not pregnant as confirmed by negative serum pregnancy test at time of screening, and is practicing one of the following methods of birth control: oral or parenteral contraceptives for three months prior to study drug administration, a vasectomized partner, or abstinence from sexual intercourse.
3. Subject is initially intubated and mechanically ventilated, or is planned for imminent intubation and mechanical ventilation, sedation is anticipated to be required during mechanical ventilation, and mechanical ventilation is anticipated to continue for at least 72 hours.
4. Subject or subject's legally authorized representative has voluntarily signed and dated an informed consent form, approved by the applicable Institutional Review Board (IRB), after the nature of the study has been explained and the subject or subject's legally authorized representative has had the opportunity to ask questions. The informed consent must be signed before any study specific procedures are performed.
5. Subject is sedated within a Richmond Agitation-Sedation Scale (RASS) range of -2 to +1 at the time of initiation of study drug

Exclusion Criteria:

1. Subject has been intubated for greater than 96 hours prior to the initiation of study drug (thus, the attainment of consent, screening evaluations, and randomization must all have been completed by the 96th hour post-intubation, so that the actual initiation of the study drug infusion may start by the end of the 96 hour window).
2. Subject has serious central nervous system pathology/trauma that, per clinical judgment of the Investigator, precludes responsiveness or survival.
3. Subject for whom opiates, benzodiazepines, or dexmedetomidine are contraindicated, or who has known or suspected serious allergy to any drug that might be administered during the course of the study.
4. Subject for whom alpha-2 agonists are contraindicated.
5. Subject requires neuromuscular blocking agents during the study for use other than intubation.
6. Subject requires epidural or spinal analgesia during the study.
7. Subject meets any of the following cardiovascular criteria:

   * Acute unstable angina (defined during current hospital stay).
   * Suspicion of acute myocardial infarction.
   * Considered to have a left ventricular ejection fraction of less than 30%. Decision to exclude is predicated on the Investigator's opinion, and may be based on any combination of acute presentations, recently performed diagnostic studies, or a history that suggests poor cardiac function. Pulmonary congestion of a non-cardiac origin or mild congestive failure primarily attributable to etiologies other than poor ventricular function are not exclusion criteria.
   * Heart rate <50 bpm prior to infusion start.
   * Systolic blood pressure <90 mmHg prior to infusion start.
   * Conduction abnormalities except 1st degree AV block and rate-controlled atrial fibrillation; subjects with functional pacemaker capacity may be enrolled.
8. Subject is hospitalized primarily due to trauma and/or burns, has received general anaesthesia within the 24 hours prior to the start of study drug infusion, or is anticipated to require general anaesthesia within 24 hours after the start of the infusion.
9. Subject has participated in a trial with any experimental drug within 30 days prior to enrollment in the study, or has ever been enrolled in this study.
10. Subject is unable to undergo any procedure required by the protocol.
11. Subject has laboratory results indicating the presence of liver disease consistent with a Child-Pugh score >9 (Grade C).
12. Subject has acute hepatitis, history or presence of chronic hepatitis, and/or has had a positive result for Hepatitis B Surface Antigen Test.
13. Subject requires dialysis (eg, hemodialysis, peritoneal dialysis, Continuous Venovenous Hemodialysis [CVVHD]).
14. Subject has a known, uncontrolled seizure disorder.
15. Subject has, per the Investigator's judgment, a known or suspected physical or psychological dependence on an abused drug, other than alcohol.
16. Subject has a known psychiatric illness that could confound a normal response to sedative treatment.
17. Subject is incarcerated.
18. Subject is terminally ill with a life duration expectancy of ≤60 days.
19. Subject has any other condition or factor which, in the Investigator's opinion, might increase the risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2005-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The percentage of time spent within the protocol specified sedation range (Richmond Agitation-Sedation Scale [RASS] range of -2 to +1) | Preinfusion, Treatment period: every 10min for 30min, 1 & 4 hr after infusion starts, every 4 hrs, prior to end of infusion & extubation. Follow-up Period (48hrs): every 10min for 1st 30min after drug discontinuation, 1, 4, 8,12, 24 & 48 hr post infusion
  RASS Range:
  Score +1 (Restless: Anxious; but movements not aggressive or vigorous) Score 0 (Alert and calm) Score -1 (Drowsy: Not fully alert, but has sustained awakening [eye opening/eye contact] to voice [≥10 seconds]) Score -2 (Light sedation: Briefly awakens with eye contact to voice [< 10 seconds])

SECONDARY OUTCOMES:
Percentage of subjects able to achieve a RASS between - 2 and +1 without interruption of study drug | Preinfusion, Treatment period: every 10min for 30min, 1 & 4 hr after infusion starts, every 4 hrs, prior to end of infusion & extubation. Follow-up Period (48hrs): every 10min for 1st 30min after drug discontinuation, 1, 4, 8,12, 24 & 48 hr post infusion
Percentage of subjects with evidence of delirium (Confusion Assessment Method [CAM]-ICU positive) while on study drug | Prior to the start of the study drug infusion. Daily each morning beginning the day after starting study drug, and at the end of study drug infusion.
Percentage of subjects with evidence of delirium (CAM-ICU positive) following discontinuation of study drug | At 12, 24, 36, and 48 hrs after end of infusion. Every 12 hours during the 48-hour Follow-Up Period.
Time to achieving a RASS between -2 and +1 for daily arousal assessment | Prior to the start of the study drug infusion. Daily each morning beginning the day after starting study drug, and at the end of study drug infusion.
Percentage of subjects who can interact with caregivers | Prior to start of infusion (Day 0), daily each morning throughout the Treatment Period beginning on the day after randomization (Study Day 1), and immediately prior to discontinuation of study drug infusion at the end of Treatment Period.
  Percentage of subjects who can interact with caregivers (i.e., follow at least 3 of the 4 arousal assessment commands) while in the protocol-specified RASS range of -2 to +1
Overall drug (sedative) tolerance | During the treatment period (Approximately 30 days)
Fentanyl use | During the treatment period (Approximately 30 days)
Nursing assessment | Screening period, during the treatment period (Approximately 30 days), and 48-hours of follow-up period
Use of rescue midazolam for sedation | During the treatment period (Approximately 30 days)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (78):
  - Birmingham, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Rogers, Arkansas
  - Davis, California
  - Loma Linda, California
  - Palo Alto, California
  - Pasadena, California
  - Redlands, California
  - Sacramento, California
  - San Clemente, California
  - San Francisco, California
  - San Jose, California
  - Denver, Colorado
  - Farmington, Connecticut
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Bay Pines, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Gordon, Georgia
  - Arlington Heights, Illinois
  - Oak Park, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Olathe, Kansas
  - Hazard, Kentucky
  - Louisville, Kentucky
  - Alexandria, Louisiana
  - Shreveport, Louisiana
  - Biddeford, Maine
  - Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Flint, Michigan
  - Missoula, Montana
  - Omaha, Nebraska
  - Camden, New Jersey
  - Englewood, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - Stoney Brook, New York
  - Syracuse, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Dayton, Ohio
  - Kettering, Ohio
  - Toledo, Ohio
  - Olkahoma City, Oklahoma
  - Medford, Oregon
  - Danville, Pennsylvania
  - Monroeville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Spartanburg, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Ogden, Utah
  - Lynchburg, Virginia
  - Morgantown, West Virginia
  - Madison, Wisconsin
- Ciudad de Buenos Aires, Argentina
- Australia (8):
  - Blacktown, New South Wales
  - Randwick, New South Wales
  - Woodville, South Australia
  - Hobart, Tasmania
  - Box Hill, Victoria
  - Heidelberg, Victoria
  - Parkville, Victoria
  - Perth, Western Australia
- Brazil (4):
  - Porto Alegre, Rio Grande do Sul
  - Pedro de Toledo, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
- New Zealand (4):
  - Christchurch
  - Hastings
  - Palmerston North
  - Welling

REFERENCES:
- [Derived] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334